CLINICAL TRIAL: NCT03834428
Title: IText For ICOUGH: Improving Ambulation of Surgical Patients Through Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-38265
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Ambulation Difficulty
Keywords: Text message reminder; ICOUGH protocol; IText; Safety net hospital; Inpatient
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Text Message Control (Active Comparator): Participants randomized to this arm will receive education about the ICOUGH protocol which includes the importance of ambulation.
  Interventions: Behavioral: ICOUGH protocol
- Text Message Intervention (Experimental): Participants randomized to this arm will receive daily text message reminders to ambulate in the hospital in addition to education about the ICOUGH protocol which includes the importance of ambulation.
  Interventions: Behavioral: Text Message Intervention; Behavioral: ICOUGH protocol

INTERVENTIONS:
Behavioral: Text Message Intervention — A text message will be sent once daily (between noon and 3p) to remind participants to ambulate at least 3 times each day while hospitalized.
  Arms: Text Message Intervention
Behavioral: ICOUGH protocol — Education will be provided about the ICOUGH protocol which includes: Incentive spirometry (a breathing device that expands the lungs), Coughing and deep breathing, Oral hygiene (for example using a toothbrush), Understanding (patient and family education), Getting out of bed at least three times daily, and Head-of-bed elevation to prevent choking.

SUMMARY:
The investigators plan to conduct a study that evaluates if text messaging increases patients' adherence to ambulation (specifically reminding patients to get out of bed three or more times daily) which is one component of a protocol called ICOUGH, which is a mnemonic that stands for: Incentive spirometry (a breathing device that expands the lungs), Coughing and deep breathing, Oral hygiene (using a toothbrush for example),Understanding (patient and family education), Getting out of bed at least three times daily, and Head-of-bed elevation to prevent choking; each letter representing steps of a protocol developed at Boston Medical Center (BMC) shown to decrease lung-related complications of surgery. Other outcomes, including frequency of ambulation, pain score, number of visitors per day, head-of-bed elevation, education on importance of ambulation, and falls will also be assessed. The hypothesis is that a reminder text message to ambulate will improve these outcomes over time.

While beneficial to patients and health care facilities, the ICOUGH protocol is sometimes both difficult to implement and sustain at an acute care hospital, because: (1) patient motivation fluctuates and is the key determinant of patient ambulation (2) it relies heavily on nurses to both educate patients and then keep them accountable to the protocol, (3) an unfavorable nurse-to-patient ratio, (4) high inpatient turnover for elective surgical cases, and (5) an aging baby boomer population-a higher volume of older, higher- risk patients will require more time and attention per nurse. Therefore, utilization of text message reminders may promote better patient, family, and provider engagement and adherence to ambulation which can improve outcomes and decrease healthcare spending.

DETAILED DESCRIPTION:
Pulmonary complications (e.g., pneumonia, unplanned intubation, and prolonged duration of ventilatory support) occur after about 1-2% of operations in the United States, leading to significant morbidity, lengths of hospital stay and cost, perhaps as much as $50,000 in expenses for the necessary additional care. However, many of these complications are preventable and the ICOUGH protocol has been demonstrated to impact pulmonary post operative complications. It has been shown to improve patient outcomes by decreasing postoperative pneumonia by 38%, unplanned intubations by 40%, and all adverse outcomes by 40%; over $5 million in cost savings for BMC in a two-year period has accompanied improved patient outcomes.

But despite its efficacy, the acute care hospital setting, specifically a safety-net hospital setting, presents challenges to ICOUGH protocol sustainability. ICOUGH requires education of patients over a number of time points and holds them accountable to adhere to the protocol. Nurses represent one source of education, although other clinical demands compete for nurses' time and attention. Acute care hospitals face high inpatient turnover for elective operations and must contend with an aging population that translates to a higher volume of older, higher-risk patients who may require more time and attention per nurse. Additionally, non-elective surgery patients, such as those admitted from the emergency department, would not have received ICOUGH protocol education. However, patients who are admitted to the hospital after emergency and trauma operations are at greatest risk of suffering pulmonary complications and stand to benefit the most from these interventions. These patients are not always optimized for surgery due to their acute circumstances, and they do not ordinarily receive the ICOUGH education that patients have prior to elective operations. In addition, patients also lack significant motivation due to the seriousness of their presentation and pain level to ambulate unless reminded.

To address these challenges within BMC and facilitate ambulation protocol implementation, sustainability, and scaling in other institutions, the research team developed a point-of-care, patient-centric way to promote better patient, family, and provider engagement with and adherence to the ICOUGH protocol, specifically ambulation. In this pilot study, patients will be randomized to receive a text message once a day to remind them to ambulate three or more times each day in addition to the ICOUGH education or to receive the ICOUGH education without text reminders. All participants will be contacted daily by a research team member to collect data on the outcome measures and each participant in the experimental text message arm will be interviewed at hospital discharge to solicit their opinion abut the text message reminders.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders on any surgical service at Boston Medical Center
* English speaking
* Ability to read at 5th grade level
* Able to ambulate, with or without assistance
* Possession of a personal cell phone that can receive text messages

Exclusion Criteria:

* Visually impaired or blind
* Presence of neuromuscular disease or inability to perform all the measures in the ICOUGH protocol
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of ambulation daily while hospitalized | baseline and 10 days
  The frequency of ambulation will be tracked for each participant each day of their hospitalization after ICOUGH education. Ambulation is defined as leaving a patient's room.

SECONDARY OUTCOMES:
Pain Level Scale twice daily while hospitalized | Twice daily until hospital discharge or for 10 days maximum
  Participants will be asked twice daily (in the morning and evening) until discharge, "On a scale of 1-10, with 10 being the worst pain imaginable, what is your pain now?" Lower scores are more favorable.
Number of participants that received ambulation education during hospitalization | At hospital discharge or hospital day #10
  Participants will be asked whether they received any education on the importance of ambulation while hospitalized.
Daily chair usage during hospitalization | Daily until hospital discharge or for 10 days maximum
  Participants will be asked about the number of times they sit in the chair in their room each day.
Number of daily visitors while hospitalized | Daily until hospital discharge or for 10 days maximum
  Participants will be asked how many visitors they had while hospitalized
Number of visitors who helped participants ambulate | Daily until hospital discharge or for 10 days maximum
  Participants will be asked how many visitors helped them ambulate.
Usefulness of the text messages in the experimental group | At hospital discharge or hospital day #10
  At discharge participants in the experimental arm will be interviewed as to their opinions about the text messages. The qualitative answers will be analyzed for themes and content.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Rosenkranz, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No